CLINICAL TRIAL: NCT02344823
Title: Effect of Vardenafil on Erectile Dysfunction and Portal Hemodynamics in Patients With Liver Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arnulf Ferlitsch, MD, Assoz. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EUDRACT: 2010-023420-25
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Cirrhosis; Erectile Dysfunction
Keywords: cirrhosis; erectile dysfunction; portal hypertension
MeSH Terms: conditions — Fibrosis; Erectile Dysfunction; Hypertension, Portal | interventions — Vardenafil Dihydrochloride; BaseLine dental cement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vardenafil Phase A (Active Comparator): HVPG (Hepatic Venous Pressure Measurement) at baseline and Response to Vardenafil 10mg per oral for 7 days at day 7 IIEF5 at baseline and day 7
  Interventions: Drug: Vardenafil; Procedure: HVPG (Hepatic venous pressure measurement) baseline; Procedure: HVPG (Hepatic venous pressure measurement) day 7; Behavioral: IIEF 5 (International Index of Erectile Function) questionaire baseline; Behavioral: IIEF 5 (International Index of Erectile Function) questionnaire at study phase end
- Placebo Phase A (Placebo Comparator): HVPG (Hepatic Venous Pressure Measurement) Measurement at baseline and Response to Placebo per oral for 7 days at day 7 IIEF 5 at baseline and day 7
  Interventions: Procedure: HVPG (Hepatic venous pressure measurement) baseline; Procedure: HVPG (Hepatic venous pressure measurement) day 7; Behavioral: IIEF 5 (International Index of Erectile Function) questionaire baseline; Behavioral: IIEF 5 (International Index of Erectile Function) questionnaire at study phase end; Drug: Placebo intake once daily
- Vardenfil Phase B (Active Comparator): IIEF 5 (International Index of Erectile Function) at baseline and Response to Vardenafil 10mg per oral ad libidum in 28 days at day 28
  Interventions: Drug: Vardenafil; Behavioral: IIEF 5 (International Index of Erectile Function) questionaire baseline; Behavioral: IIEF 5 (International Index of Erectile Function) questionnaire at study phase end
- Placebo Phase B (Placebo Comparator): IIEF 5 (International Index of Erectile Function) at baseline and Response to Placebo per oral ad libidum in 28 days at day 28
  Interventions: Behavioral: IIEF 5 (International Index of Erectile Function) questionaire baseline; Behavioral: IIEF 5 (International Index of Erectile Function) questionnaire at study phase end; Drug: Placebo intake once daily

INTERVENTIONS:
Drug: Vardenafil — per oral intake of 10mg Vardenafil once daily
  Arms: Vardenafil Phase A; Vardenfil Phase B
Procedure: HVPG (Hepatic venous pressure measurement) baseline — HVPG measurement day 1
  Other Names: HVPG
  Arms: Placebo Phase A; Vardenafil Phase A
Procedure: HVPG (Hepatic venous pressure measurement) day 7 — HVPG measurement day 7
  Other Names: HVPG
  Arms: Placebo Phase A; Vardenafil Phase A
Behavioral: IIEF 5 (International Index of Erectile Function) questionaire baseline — IIEF 5 questionaire to define level of erectile dysfunction at baseline
  Other Names: IIEF 5
Behavioral: IIEF 5 (International Index of Erectile Function) questionnaire at study phase end — IIEF 5 questionaire to define level of erectile dysfunction at end of study phase
  Other Names: IIEF 5
Drug: Placebo intake once daily
  Arms: Placebo Phase A; Placebo Phase B

SUMMARY:
The investigators want to analyze the effect of Vardenafil on Erectile Dysfunstion and portal hemodynamics in patients with liver cirrhosis.

DETAILED DESCRIPTION:
2 Phase 2 arm study

Phase A:

Baseline HVPG (Hepatic Venous Pressure Measurement) measurement, followed by 1 capsule of 10mg Vardenafil or Placebo (randomization 1:1) daily per oral for 7 days, HVPG measurement at day 7

Phase B:

1 capsule of 10mg Vardenafil or Placebo (randomization 1:1) ad libidum per oral for 28 days

ELIGIBILITY:
Inclusion Criteria:

* Male patients aged older than 18 years with mild to moderate (Child´s Grade A or B) cirrhosis scheduled for hepatic hemodynamic investigation.
* Erectile dysfunction in medical history
* Following beta-blocker therapy will be allowed: carvedilol (up to the max. dose of 25 mg) and propranolol (up to the max. dose of 160 mg)
* Patient living in a stable relationship
* HVPG (Hepatic Venous Pressure Measurement)>= 10 mmHg

Exclusion Criteria:

* HVPG <10
* HVPG > 20 mmHg and varices, unless ligated and treated in an eradication program within 6 months
* history of variceal bleeding without secondary prophylaxis with beta blocker or endoscopic band ligation
* History of endoscopically diagnosed large varices with red spots without previous bleeding and without prophylactic beta blocker or endoscopic band ligation
* History of hypersensitivity to the trial drugs and contrast agent or to drugs with a similar chemical structure
* Treatment with vasoactive or non-steroidal anti-inflammatory drugs or systemic antibiotics one week before the study
* Exclusion criteras for hepatic hemodynamic investigation
* Cardiac, renal or respiratory failure
* previous surgical or transjugular intrahepatic portosystemic shunt
* insulin-dependent diabetes
* Child´s Grade C cirrhosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
HVPG (Hepatic Venous Pressure Measurement) | 7 days
  HVPG response to Vardenafil/Placebo at day 7
IIEF (International Index of Erectile Function ) 5 | 28 days
  IIEF 5 calculation after Vardenafil/Placebo both Phase A and B

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Internal Medicine III, Gastroenterology and Hepatology, Medical University of Vienna, Vienna, Austria